CLINICAL TRIAL: NCT03725826
Title: Risk Stratification for Sudden Cardiac Death After Acute Myocardial Infarction by Measuring Left Ventricular Volume Scar With Cardiac MRI
Brief Title: Risk Stratification After Acute Myocardial Infarction With Cardiac MRI
Acronym: CR-2280
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Mario Garcia, Professor, Montefiore Medical Center
Other Study IDs: 13-01-023
Record Dates: First submitted 2014-05-02; First posted 2018-10-31 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Acute Myocardial Infarction (AMI)
Keywords: Sudden Cardiac Death; Acute Myocardial Infarction; Implantable Cardioverter Defibrillator; Cardiac Magnetic Resonance
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute Myocardial Infarction: Patients (aged 18 and above) with either ST segment elevation or Non-ST segment elevation MI by biomarkers of cardiac injury and symptoms. Cut-off for CPK >2 times and troponin >3 times the upper limit for the lab. Only Patients who undergo coronary revascularization (PCI, CABG), New York Heart Association (NYHA) functional class I-III, and with LVEF < 45% will be enrolled.

SUMMARY:
Given the existing controversy regarding the appropriate determination time for placement of implantable cardioverter-defibrillator (ICD) in patients at risk for sudden cardiac death (SCD) following acute myocardial infarction (AMI), the modest ability of current criteria to determine which patients will experience SCD, and the high impact of SCD to society, we propose to conduct a prospective non-randomized observational study to determine:

* Whether quantification of left ventricular (LV) scar volume by cardiac magnetic resonance (CMRI) prior to hospital discharge helps to predict which patients will have a low ejection fraction (35%) at follow up and qualify for ICD implantation.
* Whether quantification of infarct scar volume by CMRI will help to identify which patients will experience malignant ventricular arrhythmias and/or SCD at follow-up, independent of the LV ejection fraction (LVEF).

Primary hypothesis:

Percentage of left ventricular scar volume as measured by CMRI post-MI strongly correlates with LVEF at 40 days and 3 months.

Secondary hypothesis:

1. A volume of >40% of left ventricular scar measured by CMRI post-MI is predictive of LVEF less than 35% at 40 days and at 3 months
2. Volume scar as measured by Cardiac magnetic resonance imaging after AMI (at day 5) is predictive of clinical outcomes: SCD, total mortality, heart failure admission and life-threatening malignant ventricular arrhythmias regardless of ejection fraction at 40 days and at 3 months.

Safety hypothesis:

ICDs will be implanted if patients meet criteria at 40 days post MI as per the current American College of Cardiology (ACC) /American Heart Association (AHA) /Heart Rhythm Society (HRS) 2008 Guidelines for Device-Based Therapy of Cardiac Rhythm Abnormalities

ELIGIBILITY:
Inclusion Criteria:

* Evidence of AMI either ST segment elevation or Non-ST segment elevation MI by biomarkers of cardiac injury and symptoms. Cut-off for creatine phosphokinase (CPK) >2 times and troponin >3 times the upper limit for the lab. Only Patients who undergo coronary revascularization (PCI, CABG) will be enrolled.
* LVEF < 45%. (Based on 10 points SD in echo measurements for LVEF)
* NYHA functional class I-III
* Patients aged 18 or above, both genders.

Exclusion Criteria:

* Patients with spontaneous or induced sustained ventricular tachycardia after 48-72 hours. (30 beats or more at 120 bpm or greater)
* Absolute contraindications to undergo CMRI (Renal failure with GFR<30% or ICD/PPM)
* Antiarrhythmic medications for ventricular arrhythmias (other than beta-blockers)
* Severe non-ischemic cardiac pathology. (e.g., ARVD, HCM, severe, restrictive cardiomyopathies (amiloydosis/sarcoidosis). We are aware that non-ischemic and ischemic cardiomyopathy may co-exist. However, these cardiomyopathies convey further arrhythmic risk and diffuse LV impairment.
* Unwilling or unable to provide informed consent
* Life expectancy less than 1 year.
* Current drug or alcohol abuse.
* Pregnancy
* Claustrophobia
* Patients who are enrolled in other trials with a treatment arm. (Patients enrolled in diagnostic trials can be included).
* Difficulty to attend the follow-up schedule due to a history of medical noncompliance, living a distance from the study center, or anticipated nonresidence in the area for the length of time required for follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The proposed clinical setting of this observational study is mainly the community served by Montefiore Medical Center, the University Hospital of Albert Einstein College of Medicine. We will recruit approximately 200 patients over a year. This study will involve our two divisions (Moses and Weiler) and each study center will enroll approximately 100 patients per year.
  AMI survivors either on telemetry floor or coronary care units who meet inclusion/exclusion criteria will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in LVEF in post MI patients | 40 days post-MI and 3 months post-MI
  The degree of LVEF recovery after a first MI provides important prognostic information. Patients with no recovery in LVEF after MI are at high risk of sudden cardiac arrest events and death.

SECONDARY OUTCOMES:
LVEF less than 35% | At 40 days post-MI
  The degree of LVEF recovery after a first MI provides important prognostic information. Patients with no recovery in LVEF after MI are at high risk of sudden cardiac arrest events and death.
Cardiovascular Mortality | At 40 days post-MI
  Cardiovascular mortality in patients was defined as death attributable to myocardial ischemia and infarction, heart failure, cardiac arrest because of other or unknown cause, or cerebrovascular accident.
Cardiovascular Mortality | at 3 months post-MI
  Cardiovascular mortality in patients was defined as death attributable to myocardial ischemia and infarction, heart failure, cardiac arrest because of other or unknown cause, or cerebrovascular accident.
Sustained ventricular tachycardia (VT) | At 40 days post-MI
  Sustained ventricular tachycardia (VT) is a ventricular rhythm faster than 100 bpm lasting at least 30 seconds or requiring termination earlier due to hemodynamic instability. VT is defined as a wide complex tachycardia (QRS 120 milliseconds or greater) that originates from one of the ventricles, and is not due to aberrant conduction (e.g., from bundle branch block), at a rate of 100 bpm or greater.
Sustained ventricular fibrillation (VF) | At 40 days post-MI
  Sustained ventricular fibrillation is malignant arrhythmia
Sustained ventricular tachycardia (VT) | At 3 months post-MI
  Sustained ventricular tachycardia (VT) is a ventricular rhythm faster than 100 bpm lasting at least 30 seconds or requiring termination earlier due to hemodynamic instability. VT is defined as a wide complex tachycardia (QRS 120 milliseconds or greater) that originates from one of the ventricles, and is not due to aberrant conduction (e.g., from bundle branch block), at a rate of 100 bpm or greater.
Sustained ventricular fibrillation (VF) | At 3 months post-MI
  Sustained ventricular fibrillation is malignant arrhythmia

OTHER OUTCOMES:
Repeated Emergency Department visits | At 40 days post-MI
  Safety outcomes include repeat Emergency Department (ED) visits, hospital admissions and major adverse cardiovascular events (all-cause mortality, cardiac death, non-fatal myocardial infarction and stroke). Performance of subsequent cardiac imaging studies, cardiac catheterization and coronary interventions will also be monitored as a reflection of test efficiency.
Hospital admissions | At 40 days post-MI
  Safety outcomes include include repeat ED visits, hospital admissions and major adverse cardiovascular events (all-cause mortality, cardiac death, non-fatal myocardial infarction and stroke). Performance of subsequent cardiac imaging studies, cardiac catheterization and coronary interventions will also be monitored as a reflection of test efficiency.
All-cause mortality | At 40 days post-MI
  Safety outcomes include include repeat ED visits, hospital admissions and major adverse cardiovascular events (all-cause mortality, cardiac death, non-fatal myocardial infarction and stroke). Performance of subsequent cardiac imaging studies, cardiac catheterization and coronary interventions will also be monitored as a reflection of test efficiency.
Cardiac death | At 40 days post-MI
  Safety outcomes include include repeat ED visits, hospital admissions and major adverse cardiovascular events (all-cause mortality, cardiac death, non-fatal myocardial infarction and stroke). Performance of subsequent cardiac imaging studies, cardiac catheterization and coronary interventions will also be monitored as a reflection of test efficiency.
non-fatal myocardial infarction | At 40 days post-MI
  Safety outcomes include include repeat ED visits, hospital admissions and major adverse cardiovascular events (all-cause mortality, cardiac death, non-fatal myocardial infarction and stroke). Performance of subsequent cardiac imaging studies, cardiac catheterization and coronary interventions will also be monitored as a reflection of test efficiency.
Incidents of Stroke | At 40 days post-MI
  Safety outcomes include include repeat ED visits, hospital admissions and major adverse cardiovascular events (all-cause mortality, cardiac death, non-fatal myocardial infarction and stroke). Performance of subsequent cardiac imaging studies, cardiac catheterization and coronary interventions will also be monitored as a reflection of test efficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Garcia, M.D., Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, Albert Einstein College of Medicine, The Bronx, New York, United States

REFERENCES:
- [Background] Zipes DP, Camm AJ, Borggrefe M, Buxton AE, Chaitman B, Fromer M, Gregoratos G, Klein G, Moss AJ, Myerburg RJ, Priori SG, Quinones MA, Roden DM, Silka MJ, Tracy C, Smith SC Jr, Jacobs AK, Adams CD, Antman EM, Anderson JL, Hunt SA, Halperin JL, Nishimura R, Ornato JP, Page RL, Riegel B, Blanc JJ, Budaj A, Dean V, Deckers JW, Despres C, Dickstein K, Lekakis J, McGregor K, Metra M, Morais J, Osterspey A, Tamargo JL, Zamorano JL; American College of Cardiology/American Heart Association Task Force; European Society of Cardiology Committee for Practice Guidelines; European Heart Rhythm Association; Heart Rhythm Society. ACC/AHA/ESC 2006 Guidelines for Management of Patients With Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death: a report of the American College of Cardiology/American Heart Association Task Force and the European Society of Cardiology Committee for Practice Guidelines (writing committee to develop Guidelines for Management of Patients With Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death): developed in collaboration with the European Heart Rhythm Association and the Heart Rhythm Society. Circulation. 2006 Sep 5;114(10):e385-484. doi: 10.1161/CIRCULATIONAHA.106.178233. Epub 2006 Aug 25. No abstract available. PMID 16935995
- [Background] Adabag AS, Therneau TM, Gersh BJ, Weston SA, Roger VL. Sudden death after myocardial infarction. JAMA. 2008 Nov 5;300(17):2022-9. doi: 10.1001/jama.2008.553. PMID 18984889
- [Background] Bailey JJ, Berson AS, Handelsman H, Hodges M. Utility of current risk stratification tests for predicting major arrhythmic events after myocardial infarction. J Am Coll Cardiol. 2001 Dec;38(7):1902-11. doi: 10.1016/s0735-1097(01)01667-9. PMID 11738292
- [Background] Epstein AE, DiMarco JP, Ellenbogen KA, Estes NA 3rd, Freedman RA, Gettes LS, Gillinov AM, Gregoratos G, Hammill SC, Hayes DL, Hlatky MA, Newby LK, Page RL, Schoenfeld MH, Silka MJ, Stevenson LW, Sweeney MO, Smith SC Jr, Jacobs AK, Adams CD, Anderson JL, Buller CE, Creager MA, Ettinger SM, Faxon DP, Halperin JL, Hiratzka LF, Hunt SA, Krumholz HM, Kushner FG, Lytle BW, Nishimura RA, Ornato JP, Page RL, Riegel B, Tarkington LG, Yancy CW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the ACC/AHA/NASPE 2002 Guideline Update for Implantation of Cardiac Pacemakers and Antiarrhythmia Devices); American Association for Thoracic Surgery; Society of Thoracic Surgeons. ACC/AHA/HRS 2008 Guidelines for Device-Based Therapy of Cardiac Rhythm Abnormalities: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the ACC/AHA/NASPE 2002 Guideline Update for Implantation of Cardiac Pacemakers and Antiarrhythmia Devices) developed in collaboration with the American Association for Thoracic Surgery and Society of Thoracic Surgeons. J Am Coll Cardiol. 2008 May 27;51(21):e1-62. doi: 10.1016/j.jacc.2008.02.032. No abstract available. PMID 18498951
- [Background] Bigger JT Jr. Prophylactic use of implanted cardiac defibrillators in patients at high risk for ventricular arrhythmias after coronary-artery bypass graft surgery. Coronary Artery Bypass Graft (CABG) Patch Trial Investigators. N Engl J Med. 1997 Nov 27;337(22):1569-75. doi: 10.1056/NEJM199711273372201. PMID 9371853
- [Background] Hohnloser SH, Kuck KH, Dorian P, Roberts RS, Hampton JR, Hatala R, Fain E, Gent M, Connolly SJ; DINAMIT Investigators. Prophylactic use of an implantable cardioverter-defibrillator after acute myocardial infarction. N Engl J Med. 2004 Dec 9;351(24):2481-8. doi: 10.1056/NEJMoa041489. PMID 15590950
- [Background] Multicenter Postinfarction Research Group. Risk stratification and survival after myocardial infarction. N Engl J Med. 1983 Aug 11;309(6):331-6. doi: 10.1056/NEJM198308113090602. PMID 6866068
- [Background] Zaret BL, Wackers FJ, Terrin ML, Forman SA, Williams DO, Knatterud GL, Braunwald E. Value of radionuclide rest and exercise left ventricular ejection fraction in assessing survival of patients after thrombolytic therapy for acute myocardial infarction: results of Thrombolysis in Myocardial Infarction (TIMI) phase II study. The TIMI Study Group. J Am Coll Cardiol. 1995 Jul;26(1):73-9. doi: 10.1016/0735-1097(95)00146-q. PMID 7797778
- [Background] Antman EM, Anbe DT, Armstrong PW, Bates ER, Green LA, Hand M, Hochman JS, Krumholz HM, Kushner FG, Lamas GA, Mullany CJ, Ornato JP, Pearle DL, Sloan MA, Smith SC Jr; American College of Cardiology; American Heart Association; Canadian Cardiovascular Society. ACC/AHA guidelines for the management of patients with ST-elevation myocardial infarction--executive summary. A report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to revise the 1999 guidelines for the management of patients with acute myocardial infarction). J Am Coll Cardiol. 2004 Aug 4;44(3):671-719. doi: 10.1016/j.jacc.2004.07.002. No abstract available. PMID 15358045
- [Background] Burns RJ, Gibbons RJ, Yi Q, Roberts RS, Miller TD, Schaer GL, Anderson JL, Yusuf S; CORE Study Investigators. The relationships of left ventricular ejection fraction, end-systolic volume index and infarct size to six-month mortality after hospital discharge following myocardial infarction treated by thrombolysis. J Am Coll Cardiol. 2002 Jan 2;39(1):30-6. doi: 10.1016/s0735-1097(01)01711-9. PMID 11755283
- [Background] Moss AJ, Hall WJ, Cannom DS, Daubert JP, Higgins SL, Klein H, Levine JH, Saksena S, Waldo AL, Wilber D, Brown MW, Heo M. Improved survival with an implanted defibrillator in patients with coronary disease at high risk for ventricular arrhythmia. Multicenter Automatic Defibrillator Implantation Trial Investigators. N Engl J Med. 1996 Dec 26;335(26):1933-40. doi: 10.1056/NEJM199612263352601. PMID 8960472
- [Background] Buxton AE, Lee KL, Fisher JD, Josephson ME, Prystowsky EN, Hafley G. A randomized study of the prevention of sudden death in patients with coronary artery disease. Multicenter Unsustained Tachycardia Trial Investigators. N Engl J Med. 1999 Dec 16;341(25):1882-90. doi: 10.1056/NEJM199912163412503. PMID 10601507
- [Background] Urena PE, Lamas GA, Mitchell G, Flaker GC, Smith SC Jr, Wackers FJ, McEwan P, Pfeffer MA. Ejection fraction by radionuclide ventriculography and contrast left ventriculogram. A tale of two techniques. SAVE Investigators. Survival and Ventricular Enlargement. J Am Coll Cardiol. 1999 Jan;33(1):180-5. doi: 10.1016/s0735-1097(98)00533-6. PMID 9935027
- [Background] Solomon SD, Glynn RJ, Greaves S, Ajani U, Rouleau JL, Menapace F, Arnold JM, Hennekens C, Pfeffer MA. Recovery of ventricular function after myocardial infarction in the reperfusion era: the healing and early afterload reducing therapy study. Ann Intern Med. 2001 Mar 20;134(6):451-8. doi: 10.7326/0003-4819-134-6-200103200-00009. PMID 11255520
- [Background] Sheehan FH, Doerr R, Schmidt WG, Bolson EL, Uebis R, von Essen R, Effert S, Dodge HT. Early recovery of left ventricular function after thrombolytic therapy for acute myocardial infarction: an important determinant of survival. J Am Coll Cardiol. 1988 Aug;12(2):289-300. doi: 10.1016/0735-1097(88)90397-x. PMID 3392324
- [Background] Ndrepepa G, Mehilli J, Martinoff S, Schwaiger M, Schomig A, Kastrati A. Evolution of left ventricular ejection fraction and its relationship to infarct size after acute myocardial infarction. J Am Coll Cardiol. 2007 Jul 10;50(2):149-56. doi: 10.1016/j.jacc.2007.03.034. Epub 2007 Jun 21. PMID 17616299
- [Background] Buxton AE, Lee KL, DiCarlo L, Gold MR, Greer GS, Prystowsky EN, O'Toole MF, Tang A, Fisher JD, Coromilas J, Talajic M, Hafley G. Electrophysiologic testing to identify patients with coronary artery disease who are at risk for sudden death. Multicenter Unsustained Tachycardia Trial Investigators. N Engl J Med. 2000 Jun 29;342(26):1937-45. doi: 10.1056/NEJM200006293422602. PMID 10874061
- [Background] Kumar S, Sivagangabalan G, Zaman S, West EB, Narayan A, Thiagalingam A, Kovoor P. Electrophysiology-guided defibrillator implantation early after ST-elevation myocardial infarction. Heart Rhythm. 2010 Nov;7(11):1589-97. doi: 10.1016/j.hrthm.2010.07.019. Epub 2010 Jul 19. PMID 20650333
- [Background] Newby KH, Thompson T, Stebbins A, Topol EJ, Califf RM, Natale A. Sustained ventricular arrhythmias in patients receiving thrombolytic therapy: incidence and outcomes. The GUSTO Investigators. Circulation. 1998 Dec 8;98(23):2567-73. doi: 10.1161/01.cir.98.23.2567. PMID 9843464
- [Background] de Bakker JM, van Capelle FJ, Janse MJ, Tasseron S, Vermeulen JT, de Jonge N, Lahpor JR. Slow conduction in the infarcted human heart. 'Zigzag' course of activation. Circulation. 1993 Sep;88(3):915-26. doi: 10.1161/01.cir.88.3.915. PMID 8353918
- [Background] Hundley WG, Meshack BM, Willett DL, Sayad DE, Lange RA, Willard JE, Landau C, Hillis LD, Peshock RM. Comparison of quantitation of left ventricular volume, ejection fraction, and cardiac output in patients with atrial fibrillation by cine magnetic resonance imaging versus invasive measurements. Am J Cardiol. 1996 Nov 15;78(10):1119-23. doi: 10.1016/s0002-9149(96)90063-6. PMID 8914874
- [Background] Marrouche NF, Verma A, Wazni O, Schweikert R, Martin DO, Saliba W, Kilicaslan F, Cummings J, Burkhardt JD, Bhargava M, Bash D, Brachmann J, Guenther J, Hao S, Beheiry S, Rossillo A, Raviele A, Themistoclakis S, Natale A. Mode of initiation and ablation of ventricular fibrillation storms in patients with ischemic cardiomyopathy. J Am Coll Cardiol. 2004 May 5;43(9):1715-20. doi: 10.1016/j.jacc.2004.03.004. PMID 15120835